CLINICAL TRIAL: NCT02792894
Title: Evaluation of Family Networks (FaNs) for Children With Developmental Disorders and Delays Program: A Cluster Randomized Control Trial
Brief Title: Family Networks (FaNs) for Children With Developmental Disorders and Delays
Acronym: FaNs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Human Development Research Foundation, Pakistan (Other)
Collaborators: Grand Challenges Canada (Other); Autism Speaks (Other); World Health Organization (Other); Benazir Bhutto Hospital, Rawalpindi (Other Government); University of Liverpool (Other)
Responsible Party: Principal Investigator, Syed Usman Hamdani, Director, Human Development Research Foundation, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 746-05
Record Dates: First submitted 2016-06-01; First posted 2016-06-08 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Neurodevelopmental Disorders; Developmental Disabilities
Keywords: cluster randomized trial; developmental delays; neurodevelopmental disorders; autism; intellectual disability; low resource settings; family volunteers
MeSH Terms: conditions — Neurodevelopmental Disorders; Developmental Disabilities; Autistic Disorder; Intellectual Disability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced Usual Care (EUC) (No Intervention): Enhanced Usual Care comprises of normal routine visits conducted by the local community health workers / Lady Health Workers (LHWs). Care is enhanced in 2 ways: (a) LHWs in the EUC arm will receive training in identifying children with developmental disorders and delays, as well as making referrals to their primary care physicians for treatment using the WHO mhGAP training program for developmental disorders and (b) The primary care physicians will receive the training in WHO mental health GAP(mhGAP) program developmental disorders module, by WHO Collaborating Center in Rawalpindi, Pakistan.
- Family Networks program (Experimental): Intervention is administered once weekly over 9-10 weeks in a group format over 3 hours per sessions. Family networks Program (FaNs) is based on WHO mhGAP module for developmental disorders and incorporates WHO Parent Skills Training program for children with developmental disorders and delays. Parents Skills Training Program includes modules on communication, play, daily living skills, managing challenging behavior, coping with stress. Intervention is provided by the family volunteers (members of community, mostly women, who have a child affected in their families).
  Interventions: Behavioral: Family networks program

INTERVENTIONS:
Behavioral: Family networks program — Intervention, Family networks Program (FaNs), is administered once weekly over 9-10 weeks in a group format over 3 hours per sessions. Family networks Program (FaNs) is based on WHO mhGAP module for developmental disorders and incorporates WHO parent skills training program for children with developmental disorders and delays. Parents Skills Training Program includes modules on communication, play, daily living skills, managing challenging behavior, coping with stress. Intervention is provided by the family volunteers (members of community, mostly women, who have a child affected in their families).
  Arms: Family Networks program

SUMMARY:
Over 6% of children in Pakistan suffer from a developmental disorder (intellectual disability or Autistic spectrum disorder) and most receive no intervention.In an earlier proof of concept study, the investigators integrated social, technological and business innovations to develop and successfully pilot a sustainable service for such children in one rural population of 30,000. Affected families were identified through a mobile phone-based interactive voice response system, and organised into family networks. 'Champion' family volunteers were trained in evidence-based interventions. A Tablet-based android application was developed for training, monitoring and supervision of the champions, based on the World Health Organization's guidelines. The champions delivered the intervention to other families in the network. The project was sustainable and demonstrated significant improvements in the lives of children and their families in the first 6 months of its operation. The investigators are scaling-up this intervention to a population of 1 million. The investigators aim to evaluate the effectiveness and cost effectiveness of the scaled-up programme using cluster randomized control trial nested within the scale-up study.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 2-12 years,
* Screen positive on any of the Ten Questions screen questionnaire items # 1,4,5,7,8,9,10 for developmental disorders and delays.
* Developmental disorder and delay present according to clinical assessment (History & clinical examination for developmental delay in motor, communication, social, cognitive, daily living skills domains according to mhGAP developmental disorders guidelines for clinical assessment

Exclusion Criteria:

* Co-morbid physical or mental conditions in the child requiring inpatient hospitalization
* Deafness or blindness in the child
* Primary caregiver not available or unwilling to participate in the intervention program for 6 months
* Physical or mental conditions in the primary caregiver needing inpatient hospitalization or frequent outpatient visits (more than two times a month)
* Written consent not obtained for participation in the trial by the primary caregiver

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 540 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Developmental Disorders- Children Disability Assessment Schedule (DD-CDAS) | Change in DD-CDAS score at 6 months post-intervention
  The DD-CDAS is a 36-item questionnaire measuring functioning and disability. The 36 items are rated on a five-point Likert scale (1=none to 5=extreme/cannot do). The items represent cognition, mobility, self-care, getting along with others, life activities, and participation in the society. The raw scores are sum across all the items of each domain and all 36 items for a tool. Domain and total raw scores are transformed into a range from 0 to 100. The tool has been validated for children with developmental disorders in Pakistan (DD-CDAS) by our group (Hamdani et al, 2020).

SECONDARY OUTCOMES:
Caregiver-Child Interaction | Baseline (Pre treatment) and follow-up (6 months post-intervention)
  Fifteen minutes video will be recorded to capture caregiver-child interaction. Caregivers will be asked to try home routines involving the child (e.g. feeding the child, performing domestic chores) or play based routines (e.g. playing with toys or reading a book) with their child. Caregiver's facilitators and interrupters (including child's engagement and distress during social communication) and joint engagement will be rated.
Strengths and Difficulties Questionnaire (SDQ) | Baseline (Pre treatment) and follow up (6 months post-intervention)
  Parent rated, 25 items scale. Items are distributed over 5 domains: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior. Each item is rated on a 3-point Likert scale (0 = not true, 1 = somewhat true, 2 = certainly true). Total difficulty score is calculated by adding all the domain scores except prosocial problems.
Family Empowerment Scale (FES) | Baseline (Pre treatment) and follow up (6 months post-intervention)
  Parent rated, 34 items scale, consisting of 3 subscales: The family subscale (12 items) refers to the parents' management of everyday situations. The service system subscale (12 items) refers to parents' acting to obtain services to meet the child's needs. The community subscale (10 items) refers to parents' advocacy for improving services for children in general. Each item is rated on a 5-point Likert scale (1 = not true at all to 5 = very true). Scores are summed across all items for each subscale with higher scores indicating relatively more empowerment.
Inventory of Stigmatizing Experiences (Family version) | Baseline (Pre treatment) and follow up (6 months post-intervention)
  Interview-based measure of the extent of stigma faced by family. Seven items, each item is rated on a 5-point Likert scale (1 = never to 5 = always). The responses are recoded into a binary variable with 1 reflecting presence of stigma and 0 reflecting absence of stigma. Scores are summed across all items with a maximum score of 7, with lower scores indicating relatively less stigma.
Pediatric Quality of Life (PedsQL) family impact module | Baseline (Pre treatment) and follow up (6 months post-intervention)
  The 36-item PedsQL™ Family Impact Module Scales encompass 6 sub-scales measuring parent self-reported functioning: 1) Physical Functioning (6 items), 2) Emotional Functioning (5 items), 3) Social Functioning (4 items), 4) Cognitive Functioning (5 items), 5) Communication (3 items), 6) Worry (5 items), and 2 scales measuring parent-reported family functioning; 7) Daily Activities (3 items) and 8) Family Relationships (5 items). Items are rated on a 5 point Likert scale (0 never to 4 almost always). For ease of interpretability, items are reversed scored and linearly transformed to a 0-100 scale, so that higher scores indicate better HRQOL (Health-Related Quality of Life).
Client Services Receipt Inventory (CSRI) | Baseline (Pre treatment) and follow up (6 months post-intervention)
  Client Services Receipt Inventory has been adapted for use in children and families with developmental disorders.
Clinical Global Impression (CGI) | Baseline (Pre treatment) and follow up (6 months post-intervention)
  Clinical global impression (CGI) measures severity of challenges in social communication (rated from 1-7) (b) improvement in social communication at 6 months follow up (rated from 1-7). The CGI will be rated from the CCX videotapes by observers blinded to intervention allocation.

CONTACTS AND LOCATIONS:
Overall Officials: Atif Rahman, PhD, Study Director — University of Liverpool
Locations (1):
- Human Development Research Foundation, Gujar Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamdani SU, Minhas FA, Iqbal Z, Rahman A. Model for Service Delivery for Developmental Disorders in Low-Income Countries. Pediatrics. 2015 Dec;136(6):1166-72. doi: 10.1542/peds.2015-0861. PMID 26598452
- [Background] Hamdani SU, Atif N, Tariq M, Minhas FA, Iqbal Z, Rahman A. Family networks to improve outcomes in children with intellectual and developmental disorders: a qualitative study. Int J Ment Health Syst. 2014 Feb 1;8(1):7. doi: 10.1186/1752-4458-8-7. PMID 24485093
- [Background] Hamdani SU, Huma ZE, Wissow L, Rahman A, Gladstone M. Measuring functional disability in children with developmental disorders in low-resource settings: validation of Developmental Disorders-Children Disability Assessment Schedule (DD-CDAS) in rural Pakistan. Glob Ment Health (Camb). 2020 Jul 13;7:e17. doi: 10.1017/gmh.2020.10. eCollection 2020. PMID 32913656
- [Background] Hamdani SU, Akhtar P, Zill-E-Huma, Nazir H, Minhas FA, Sikander S, Wang D, Servilli C, Rahman A. WHO Parents Skills Training (PST) programme for children with developmental disorders and delays delivered by Family Volunteers in rural Pakistan: study protocol for effectiveness implementation hybrid cluster randomized controlled trial. Glob Ment Health (Camb). 2017 Jun 13;4:e11. doi: 10.1017/gmh.2017.7. eCollection 2017. PMID 29230307
- [Derived] Hamdani SU, Huma ZE, Suleman N, Akhtar P, Nazir H, Masood A, Tariq M, Koukab A, Salomone E, Pacione L, Brown F, Shire S, Sikander S, Servili C, Wang D, Minhas FA, Rahman A. Effectiveness of a technology-assisted, family volunteers delivered, brief, multicomponent parents' skills training intervention for children with developmental disorders in rural Pakistan: a cluster randomized controlled trial. Int J Ment Health Syst. 2021 May 31;15(1):53. doi: 10.1186/s13033-021-00476-w. PMID 34059074